CLINICAL TRIAL: NCT03150550
Title: Study of Mindfulness Practice Efficacy in Alcoholic Relapse Prevention
Acronym: Mindfulness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Lundbeck SAS 37-45 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-321; 2016-A00048-43 (Other: 2016-A00048-43)
Record Dates: First submitted 2017-05-04; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Alcohol Use Disorder
Keywords: Mindfulness; Alcohol; Alcohol Use Disorder; Relapse; Relapse Prevention; Cognitive-behavioral therapy
MeSH Terms: conditions — Alcoholism; Recurrence | interventions — Secondary Prevention

STUDY DESIGN:
Masking Description: Simple Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relapse Prevention (Experimental): Each patient will perform 12 classic psychotherapeutic sessions over a period of 6 weeks.
  Interventions: Behavioral: Relapse prevention
- Mindfulness Practice (Experimental): Each patient will perform 12 mindfulness psychotherapeutic sessions over a period of 6 weeks.
  Interventions: Behavioral: Mindfulness practice

INTERVENTIONS:
Behavioral: Mindfulness practice — Mindfulness interventions are behavioral cognitive psychotherapies which allow patient to identify, pay attention and accept external (sensory stimuli) and internal (cognition and emotions) phenomena.
  Arms: Mindfulness Practice
Behavioral: Relapse prevention — It's a conventional relapse prevention program which allow to measure the alcoholic relapse in the first glass consumed.
  Arms: Relapse Prevention

SUMMARY:
Among behavioral cognitive psychotherapies, new "Mindfulness" interventions allow patient to identify, pay attention and accept external (sensory stimuli) and internal (cognition and emotions) phenomena. This "to do with" training has yielded promising results in stress management, prevention of depressive relapse, management of craving and an increase in self-efficacy. Few studies (none in France) have attempted to measure the efficacy of this technique on alcohol relapse, in particular by comparing it with a usual management strategy (conventional relapse prevention therapy).

The main objective of this study is to compare the efficacy on alcoholic relapse (measured in the "first glass" consumed), from a Mindfulness therapeutic program to a conventional Relapse Prevention program. Secondary objectives are to demonstrate the efficacy of this program on craving, self-efficacy, and secondary endpoints of relapse (massive alcoholism, number of alcoholisation days).

DETAILED DESCRIPTION:
Each patient will perform 12 psychotherapeutic sessions (Mindfulness or Relapse Prevention) over a period of 6 weeks. Patients will be evaluated by a practitioner different from the practitioner who makes the psychotherapeutic management.

Patients will be assessed at inclusion (Initial visit), after the 12 sessions of management (M0), 1 month (M1), 2 month (M2), 3 month (M3), 4 month (M4), 5 month (M5), 6 month (M6), after initial visit as follows

Initial Visit

* Signature of an informed consent form.
* Demographic characteristics (gender, age, family status, professional status, level of education …)
* Clinical data (patient status, ongoing pharmacological treatment, withdrawal, previous CBT ...)
* Criteria and severity of alcohol dependence (DSM 5)
* Evaluation of depressive symptomatology and severity (HAM-D)
* Level of pre-intervention alcohol consumption (AUDIT-C)
* "Binge drinking" consumption
* Craving before alcohol withdrawal (EVA craving)
* Mindfulness Skills (KIMS)
* Self-efficacy to remain abstinent (QAE-Alcohol)
* Drinking habits (QHPBA)

After the 12 sessions (M0)

* Data on treatments in progress or change in treatment
* Depressive symptomatology and severity (HAM-D)
* Level of alcohol consumption in post-intervention (AUDIT-C)
* "Binge drinking" consumption
* Craving after alcohol withdrawal (EVA craving)
* Mindfulness Skills (KIMS)
* Self-efficacy to remain abstinent (QAE-Alcohol)
* Distribution of the 1st Daily Alcohol Logbook (TLFB)

At 1 month (M1)

* Return of the 1st Daily Alcohol Logbook (TLFB)
* Data on treatments in progress or change in treatment
* Mindfulness Skills (KIMS)
* "Binge drinking" consumption
* Self-efficacy to remain abstinent (QAE-Alcohol)
* Distribution of the 2nd Daily Alcohol Logbook (TLFB)

At 2 month (M2)

* Return of the 2nd Daily Alcohol Logbook (TLFB)
* Data on treatments in progress or change in treatment
* Mindfulness Skills (KIMS)
* "Binge drinking" consumption
* Self-efficacy to remain abstinent (QAE-Alcohol)
* Distribution of the 3th Daily Alcohol Logbook (TLFB)

At 3 month (M3)

* Return of the 3th Daily Alcohol Logbook (TLFB)
* Data on treatments in progress or change in treatment
* Mindfulness Skills (KIMS)
* "Binge drinking" consumption
* Self-efficacy to remain abstinent (QAE-Alcohol)
* Distribution of the 4th Daily Alcohol Logbook (TLFB)

At 4 month (M4)

* Return of the 4th Daily Alcohol Logbook (TLFB)
* Data on treatments in progress or change in treatment
* Mindfulness Skills (KIMS)
* "Binge drinking" consumption
* Self-efficacy to remain abstinent (QAE-Alcohol)
* Distribution of the 5th Daily Alcohol Logbook (TLFB)

At 5 month (M5)

* Return of the 5th Daily Alcohol Logbook (TLFB)
* Data on treatments in progress or change in treatment
* Mindfulness Skills (KIMS)
* "Binge drinking" consumption
* Self-efficacy to remain abstinent (QAE-Alcohol)
* Distribution of the 6th Daily Alcohol Logbook (TLFB)

At 6 month (M6)

* Return of the 6th Daily Alcohol Logbook (TLFB)
* Data on treatments in progress or change in treatment
* Mindfulness Skills (KIMS)
* "Binge drinking" consumption
* Self-efficacy to remain abstinent (QAE-Alcohol)

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 75 (including landmarks)
* Patients in withdrawal for alcohol dependence according to DSM IV criteria (1994); hospital or outpatient withdrawal of more than 10 days and less than 10 weeks.

Exclusion Criteria:

* Psychiatric comorbidity (dipsomaniac alcoholism, anteriority of one or more hypomanic or manic episodes, psychoses, severe depression, severe suicidal risk)
* Other addiction syndrome than tobacco and alcohol
* Problems that impede participation in a group, such as severe borderline personality disorder; antisocial personality; tendency to dissociation; phobias of interceptive type (panic attacks and hypochondria ...)
* Problems preventing the completion of questionnaires, such as cognitive dysfunctions, dysfunctions of attention and concentration skills, or a language barrier
* Severe recurring pathology
* Need for individual weekly follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01-21 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Number of alcoholic relapses | 6 month
  Proportion of patients with an alcohol consumption of at least one glass of alcohol

SECONDARY OUTCOMES:
Alcohol relapse time | 6 month
  Measurement : Number of days elapsed between the end of treatment and the first relapse compare between the two interventions (classic or "mindfulness")
Delay in "heavy drinking" relapse | 6 month
  Measurement : Number of days elapsed between the end of treatment and the first heavy drinking (≥4 glasses of alcohol for women and ≥6 glasses of alcohol for men) compare between the two interventions (classic or "mindfulness")
Frequency of consumption | 6 month
  Measurement : Number of consumption days during 6 month compare between the two interventions (classic or "mindfulness")
Daily quantities consumed | 6 month
  Measurement : Number of standard glasses consumed per day during 6 month compare between the two interventions (classic or "mindfulness")
Degree of mindfulness skills | 6 month
  Measurement : Score at the KIMS Scale (Kentucky Inventory of Mindfulness Skills) evaluated each month, compare before and after intervention (classic or "mindfulness")
Severity of alcohol craving | 6 month
  Measurement: Assessed daily on a VAS craving (Visual analogue scale) in the daily observation book, compare before and after intervention (classic or "mindfulness")
Level of self-efficacy | 6 month
  Measurement: Assessed daily on a VAS self-efficacy (Visual analogue scale) in the daily observation book, compare before and after intervention (classic or "mindfulness")

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, France, France